CLINICAL TRIAL: NCT05348226
Title: Effect of Sacubitril/Valsartan (ENtresto) on Left Ventricular Reverse Remodelling as Demonstrated by Cardiac Magnetic Resonance (CMR) Imaging
Brief Title: The ENVI Study: Effect of Entresto on Left Ventricular Remodelling on Cardiac MRI
Acronym: ENVI
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CAR0589
Record Dates: First submitted 2022-04-05; First posted 2022-04-27 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Cardiac Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Additional Cardiac Magnetic Resonance Scan — Standard of care medical treatment with sacubitril/valsartan (Entresto). Additional Cardiac Magnetic Resonance Imaging (CMR) Scan after 4-6 months of treatment.

SUMMARY:
A prospective, single centre, observational cohort study at University Hospital Southampton NHS Foundation Trust of 50 consecutive patients with Heart Failure with reduced Ejection Fraction and Ejection Fraction ≤35% who are eligible for sacubitril/valsartan (Entresto) initiation as per European Society of Cardiology guidelines.

Participants will have baseline and repeat cardiac magnetic resonance imaging (CMR) scans after 4-6 months of Entresto therapy. The CMR scans will be compared.

Clinical outcomes at 6 months including combined outcome of death and/or heart failure hospitalisation, KCCQ-12 questionnaire, 6-minute walk test, routine blood tests and NTproBNP will also be described.

This study will be the first to examine the effects of sacubitril/valsartan (Entresto) therapy on left ventricular reverse remodelling in patients with symptomatic HFrEF as demonstrated by Cardiac Magnetic Resonance Imaging.

DETAILED DESCRIPTION:
The landmark trial PARADIGM-HF (2014) showed that a new drug sacubitril/valsartan (Entresto) was superior to a well-established drug (ACE-Inhibitors) for patients with severe heart failure. Entresto resulted in a 20% reduction in risk of death and hospitalisations, as well as improving quality of life and symptoms. This represented a major breakthrough in heart failure treatment and guidelines changed to recommend Entresto for patients in whom heart function had not improved on conventional heart failure drug treatments.

At the same point as recommending Entresto, international heart failure guidelines also recommend an Implantable Cardioverter-Defibrillator (ICD). An ICD is a device which can detect and treat potentially life-threatening heart rhythm abnormalities, which may occur in patients with persistently severe heart failure. The risk of complications associated with ICD implantation is not insignificant, up to 15%. Currently, there is a lack of consensus between clinicians regarding when best to offer ICD implantation in relation to Entresto treatment.

The exact mechanism of how Entresto achieves its beneficial effect is not fully understood. There are studies describing an improvement in heart function on Echocardiography (ultrasound). Some studies suggest a reduction in abnormal heart rhythms. There are however, no studies describing the effects of Entresto on heart tissue or function described on Cardiac Magnetic Resonance (CMR) Imaging. CMR is a specialised non-invasive scan which is excellent at looking at characteristics of heart tissue and is the gold standard for calculating heart function.

The study will enrol 50 patients who have been referred for Entresto treatment. Participants will undergo a baseline CMR to evaluate heart characteristics and function before being started on Entresto. After 6 months, participants will receive another CMR and the two scans will be compared for differences in heart size, function and tissue characteristics.

The Investigators hypothesize that there will be an improvement in a variety of CMR parameters and the findings will help better understand the mechanisms by which this is achieved e.g. reduction in fibrosis (subtle scarring) of heart tissue. The Investigators also believe a proportion of patients will avoid the need for an ICD, due to improvement in heart function.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* HFrEF EF ≤35% despite optimisation of ACE-Inhibitor, Beta Blocker & Mineralocorticoid Receptor Antagonist and referred for Entresto initiation
* Symptomatic NYHA II-III
* Able and willing to provide informed consent
* Able to undergo Cardiac Magnetic Resonance Imaging (CMR) scan

Exclusion Criteria:

* Pre-existing cardiac device (i.e. pacemaker/defibrillator)
* Symptomatic hypotension (BP <95mmHg) - [PARADIGM exclusion]
* Severe renal failure (GFR <30)
* Hyperkalaemia (K >5.4mmol/L)
* History of angioedema
* Diagnosis of amyloidosis, sarcoidosis or HCM
* Myocardial infarction or revascularisation within the last 40 days
* Valve disease expected to require surgery
* Life expectancy <2 years secondary to any other cause (i.e. malignancy)
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic severe Heart Failure with reduced Ejection Fraction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Volume quantified on Cardiac Magnetic Resonance Imaging | 6 months
  Left ventricular Volume quantified in (ml)
Indexed Left Ventricular Volume quantified on Cardiac Magnetic Resonance Imaging | 6 months
  Weight and Height will be combined to calculate Body Surface Area (m2). Left Ventricular Volume in (ml) will be divided by Body Surface Area to give indexed value (ml/m2)
Ejection Fraction quantified on Cardiac Magnetic Resonance Imaging | 6 months
  Ejection Fraction quoted in (%)

SECONDARY OUTCOMES:
Cardiac Fibrosis quantification as measured by T1 mapping on Cardiac Magnetic Resonance Imaging | 6 months
Strain Analysis as measured by feature tracking on Cardiac Magnetic Resonance Imaging | 6 months

OTHER OUTCOMES:
Combined outcome of death and/or heart failure hospitalisation | 6 months
Quality of Life assessment: KCCQ-12 questionnaire | 6 months
  Kansas City Cardiomyopathy Questionnaire.
Quality of Life assessment: 6 Minute Walk Test | 6 months
  Distance walked (m) in 6 minutes
N-terminal pro B type natriuretic peptide (NTproBNP) | 6 months
  Blood Test

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Flett, MBBS BSc MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
TBC

REFERENCES:
- [Derived] Zheng A, Adam R, Peebles C, Harden S, Shambrook J, Abbas A, Vedwan K, Adam G, Haydock P, Cowburn P, Young C, Long J, Walkden M, Smith S, Greenwood E, Olden P, Flett A. Effect of optimisation to contemporary HFrEF medical therapy with sacubitril/valsartan (Entresto) and dapaglifloziN on left Ventricular reverse remodelling as demonstrated by cardiac magnetic resonance (CMR) Imaging: the ENVI study. Open Heart. 2024 Dec 2;11(2):e002933. doi: 10.1136/openhrt-2024-002933. PMID 39622578